CLINICAL TRIAL: NCT06748495
Title: Real-world First-line Serplulimab-based Immunochemotherapy for Extensive-stage Small Cell Lung Cancer: the Multicenter ASTRUM-005R Study
Brief Title: Real-world First-line Serplulimab-based Immunochemotherapy for Extensive-stage Small Cell Lung Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ASTRUM-005R
Record Dates: First submitted 2024-11-27; First posted 2024-12-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-11

CONDITIONS: Extensive-stage Small Cell Lung Cancer (ES-SCLC)
Keywords: Real Word
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (1):
- Serplulimab: the combination of Serplulimab and chemotherapy regimen

SUMMARY:
The phase III ASTRUM-005 study (NCT04063163) has demonstrated promising antitumor efficacy and well tolerability of first-line serplulimab combined with chemotherapy in patients with extensive-stage small cell lung cancer (ES-SCLC). However, due to the strict eligibility criteria of randomized controlled trials (RCTs), real-world data on patients with more complex and varied conditions are currently lacking. This highlights the urgent need for real-world evidence to better understand the practical effectiveness and safety of treatments. ASTRUM-005R is a multicenter real-world study conducted in China, designed to evaluate the efficacy and safety of the first-line treatment serplulimab-based immunochemotherapy for ES-SCLC in real-world clinical practice. Additionally, it aims to compare its findings with the data of the randomized controlled phase III ASTRUM-005 trial (descriptive), providing insights into optimal treatment strategies for this patient population.

DETAILED DESCRIPTION:
Lung cancer is one of the malignant tumors with the highest morbidity and mortality in the world, and can be divided into non-small cell lung cancer (NSCLC) and small cell lung cancer (SCLC) according to it's pathological type (1). SCLC is the most malignant and prone type of lung cancer, accounting for about 15% to 20% of the incidence of lung cancer, approximately 70% of SCLC patients have distant metastasis at the time of diagnosis, and the 5-year survival rate of patients with extensive-stage small cell lung cancer (ES-SCLC) is less than 1% [2-3]. The treatment of SCLC has been poor for the past 30 years, and overall survival has always been around 1 year, which is in stark contrast to the great progress in NSCLC. Until recent years, immunotherapy has brought hope to SCLC patients.

The IMpower133 trial showed that first-line treatment of ES-SCLC with atezolizumab in combination with EC regimen significantly improved PFS compared with standard chemotherapy, prolonging OS by nearly 1 month with the median OS of 12.3 months, and reducing the risk of death by 30% compared with standard chemotherapy [4]. In the CASPIAN study, which compared the efficacy and safety of durvalumab plus EP chemotherapy and EP chemotherapy alone as first-line treatment for ES-SCLC, durvalumab resulted in a sustained and clinically meaningful improvement in OS in ES-SCLC patients after more than 2 years of median follow-up, and the final analysis showed that the durvalumab plus chemotherapy arm had a median OS of 12.9 months and a 25% reduction in the risk of death compared with the chemotherapy alone arm (HR 0.75; 95% CI 0.62 0.91; P 0.0032) [5]. Based on the results of the two studies, atezolizumab in combination with chemotherapy and durvalumab in combination with chemotherapy were approved by the FDA and NMPA, respectively, for the first-line treatment of extensive-stage small cell lung cancer, from which immunotherapy established a new first-line treatment standard for extensive-stage small cell lung cancer.

Serplulimab, a recombinant anti-PD-1 humanized monoclonal antibody. The interim analysis results of the phase III clinical study (ASTRUM-005) of the first-line treatment of extensive-stage small cell lung cancer with the combination of Serplulimab and chemotherapy have been published in the top international journal JAMA. The study results showed that the combination of Serplulimab and chemotherapy could prolong OS in both the overall population and the Chinese subgroup population. The median OS of the overall population in the Serplulimab group was 15.4 months, nearly 4.5 months of survival compared with the control group. The risk of death of the overall population reduced by 38%, showing good efficacy and safety [6]. In December 2022, ESMO Asia updated the final analysis results with a median follow-up time of 19.8 months. The updated data showed that the median OS in the Serplulimab plus chemotherapy group in the intent-to-treat (ITT) population was significantly prolonged by 4.7 months and reached 15.8 months compared with the control group, reducing the risk of death by 38%, and the median OS in the Asian population was prolonged by 4.8 months and reached 15.9 months. The results of this study are the first to confirm that PD-1 inhibitors can also bring survival benefit to extensive-stage small cell lung cancer patients and enhance the confidence of immunotherapy for small cell lung cancer. At the same time, this study has also been internationally recognized. On 07 Apr 2022, FDA awarded the title of orphan drug for Serplulimab for the treatment of small cell lung cancer. On 17 Jan 2023, the combination of Serplulimab and chemotherapy was approved by China Food and Drug Administration for the first-line treatment of extensive-stage small cell lung cancer.

However, there are no real-world studies of Serplulimab in patients with extensive-stage SCLC, and clinical studies are still needed to provide evidence-based evidence.

Therefore, this multi-center, observational, real-world study aims to evaluate the efficacy and safety of first-line serplulimab-based immunochemotherapy for extensive-stage small cell lung cancer across 14 study sites from 2022 to 2024. The study assesses patient baseline characteristics, treatment regimens, and clinical outcomes to provide insights into the real-world effectiveness and safety profile of this treatment approach.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically/cytologically confirmed small cell lung cancer with staging that confirming disease stage as extensive (according to the modified American Veterans Administration Lung Cancer Society [VALG] staging system);
2. No prior systemic therapy for the diagnosis of ES-SCLC;
3. Patients previously treated with chemoradiation for limited-stage SCLC: must be treatment with curative intent and have a treatment-free interval of at least 6 months between the last dose of chemotherapy/last course, end of thoracic radiotherapy or chemoradiation and confirmation of ES-SCLC;
4. At least two cycles of treatment with Serplulimab in combination with chemotherapy with one or more documented efficacy assessments ;
5. Local radiotherapy is allowed for patients indicated for radiotherapy, including but not limited to thoracic radiotherapy, brain radiotherapy.

Exclusion Criteria:

1. Incomplete clinical information, such as no disease course, pathological diagnosis, treatment and observation of outcome data;
2. Patients with SCLC and other malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically/cytologically confirmed small cell lung cancer with staging that confirming disease stage as extensive (according to the modified American Veterans Administration Lung Cancer Society [VALG] staging system). No prior systemic therapy for the diagnosis of ES-SCLC.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-06-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 1yaer
  defined as the time from the start of chemotherapy to the first occurrence of disease progression or death due to any cause, assessed by the physician according to RECIST 1.1, with the response assessment record as the determination standard

SECONDARY OUTCOMES:
Overall survival (OS) | 1yaer
  defined as the time from the start of chemotherapy to death from any cause, assessed for patients who did not die on the study end date or the last visit date available in the database, whichever occurred first
Objective response rate (ORR) | 1yaer
  defined as the proportion of patients achieving complete response (CR) or partial response (PR) in all patients. According to RECIST 1.1 evaluation criteria, physicians use the efficacy evaluation record as the determination criteria
AEs | 1yaer
  incidence of Grade 3 and higher AEs, incidence of immune-related AEs (irAEs) (based on CTCAE 5.0 criteria)

CONTACTS AND LOCATIONS:
Overall Officials: LIN Wu, Study Chair — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No